CLINICAL TRIAL: NCT00348036
Title: Trauma Interventions for Low-income Women in Primary Care
Brief Title: Group Intervention for Interpersonal Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P20MH068450 (NIH); P20MH068450 (NIH); DSIR 83-ATAS
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2013-04-30 (Estimated); Status verified 2013-04

CONDITIONS: Post-Traumatic Stress Disorder; Depression
Keywords: Major Depression; Trauma; Primary Care; Low-Income Patients
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Depressive Disorder, Major; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group therapy (Experimental): Participants will receive interpersonal group therapy.
  Interventions: Behavioral: Group Intervention for Interpersonal Trauma
- Control (Active Comparator): Participants will receive information only on PTSD.
  Interventions: Other: Information only

INTERVENTIONS:
Behavioral: Group Intervention for Interpersonal Trauma — Participants will receive information about PTSD and depression, in the form of a brochures and a DVD about trauma and its emotional consequences. Groups will be comprised of three components at each meeting: psycho-education, current relationship issues, and coping skills. Each group session will focus on a different aspect of education. Next, relationship difficulties typically associated with the symptoms discussed in that module will be addressed, and there will be group discussion about participants' relationship difficulties. Each group will end with the therapist teaching a coping skill that fits with the issues discussed earlier.
  Arms: Group therapy
Other: Information only — Participants will receive information about PTSD and depression, in the form of a brochures and a DVD about trauma and its emotional consequences.
  Arms: Control

SUMMARY:
This study will assess the acceptability and effectiveness of a six-session, modular, repeating group for low-income women who have symptoms of depression and/or post-traumatic stress disorder following interpersonal trauma exposure.

DETAILED DESCRIPTION:
The aim of this study is to assess the acceptability and effectiveness of a six-session, modular, repeating group for low-income women who have symptoms of depression and/or post-traumatic stress disorder (PTSD) following interpersonal trauma exposure. Group participants will be recruited from public sector/safety net primary care clinics. Study participants will be randomized to immediate or delayed treatment. Participants in both conditions will receive information about PTSD and depression, in the form of a brochures and a DVD about trauma and its emotional consequences. Groups will be comprised of three components at each meeting: psycho-education, current relationship issues, and coping skills. Each group session will focus on a different aspect of education. Next, relationship difficulties typically associated with the symptoms discussed in that module will be addressed, and there will be group discussion about participants' relationship difficulties. Each group will end with the therapist teaching a coping skill that fits with the issues discussed earlier. Participants will be free to attend any of the sessions they missed during the first group when the group repeats. Participants in the delayed condition will be able to attend the groups after a 12-week waiting period. Assessments of PTSD, depression, functioning, and quality of life will be conducted at three time points: baseline (prior to the start of the group), 12 weeks after the start of the group, and 6 months from the start of the group. Gift cards will be sent to the women for completing each of the assessments.

ELIGIBILITY:
Inclusion Criteria:

* Exposure to an interpersonal traumatic event
* Diagnosis of depression or PTSD (threshold or subthreshold)
* Functional literacy

Exclusion Criteria:

* Apparent incoherence or disorientation
* Apparent intoxication at recruitment
* Hearing impairment

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-09; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
PTSD checklist | Measured at baseline, Week 12, and Month 6
Hamilton Depression Inventory | Measured at baseline, Week 12, and Month 6

SECONDARY OUTCOMES:
Inventory of Interpersonal Problems | Measured at baseline, Week 12, and Month 6
Health care utilization | Measured at baseline, Week 12, and Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie L. Green, PhD, Principal Investigator — Georgetown University Medical School Psychiatry
Locations (1):
- Georgetown University, Washington D.C., District of Columbia, United States